CLINICAL TRIAL: NCT07272759
Title: Feasibility Study of Occupation-Based 'Remediation, Education, Adaptation, Promotion' (REAP) Program Among People With Stroke in Bang
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Metropolitan University (Other)
Collaborators: Centre for the Rehabilitation of the Paralysed, Bangladesh (Other)
Responsible Party: Principal Investigator, Azharul Islam, Azharul Islam, Tokyo Metropolitan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP-ERC-R&E-0401-0479
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Educational Status; Acclimatization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke patients who are taking rehabilitation (Experimental): Stroke patients aged 18-64 years, diagnosed with stroke (ischemic/hemorrhagic) 3-6 months prior, medically stable and able to provide informed consent, MoCA score ≥18.
  Interventions: Other: Occupation-Based 'Remediation, Education, Adaptation, Promotion' (REAP) Program

INTERVENTIONS:
Other: Occupation-Based 'Remediation, Education, Adaptation, Promotion' (REAP) Program — The REAP program consists of four core components designed to address the complex needs of stroke survivors:
  1. Remediation
  2. Education
  3. Adaptation
  4. Promotion

SUMMARY:
Stroke causes major disability issues in Bangladesh and often leaves people unable to look after themselves, work, or participate in family and community life. Most stroke survivors in Bangladesh do not receive adequate rehabilitation, and existing services focus mainly on physical exercises, not on helping people return to meaningful activities.

The REAP programme is a new therapy approach that remediates skills through structured training, educates patients and families on stroke management, adapts tasks or environments to make daily activities easier, and promotes participation in meaningful roles and activities.

This study will test whether the REAP programme can be delivered successfully in a Bangladeshi rehabilitation centre, whether patients find it acceptable, and whether it helps people become more independent and improves quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64 years,
* Diagnosed with stroke (ischemic/hemorrhagic) 3-24 months prior,
* Medically stable and able to provide informed consent,
* MoCA score ≥18.

Exclusion Criteria:

* Severe receptive aphasia,
* Major psychiatric disorders,
* Unstable medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | From enrollment to 12 weeks
  Assesses independence in activities of daily living (ADLs).
Montreal Cognitive Assessment (MoCA) | Enrollment to 12 weeks
  Screens for cognitive impairment.
Bangladeshi Occupational Self-Assessment - Short Form (BOSA-SF) ( | Enrollment to 12 weeks
  Evaluates perceived occupational competence and values within the local context.
Fugl-Meyer Assessment (FMA) | Enrollment to 12 weeks
  Assesses motor recovery post-stroke
Occupational Balance Questionnaire | Enrollment to 12 weeks
  Measures balance between different occupational areas in everyday life.
Life Satisfaction Questionnaire (LiSat-11) | Enrollment to 12 weeks
  Assesses subjective life satisfaction across various domains
Zarit Caregiver Burden Scale | Enrollment to 12 weeks
  Assesses the level of burden experienced by informal caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bontje, PhD, Study Director — Tokyo Metropolitan University
Locations (1):
- Centre for the Rehabilitation of the Paralysed (CRP), Dhaka, Bangladesh